CLINICAL TRIAL: NCT04980508
Title: COVID-19 Can Cause Cavernous Smooth Muscle Damage: Investigation of the Effects of COVID-19 on Cavernous Smooth Muscle by Corpus Cavernosum Electromyography
Brief Title: Effects of COVID-19 on Cavernous Smooth Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, selman unal, Principal Investigator, Ankara Yildirim Beyazıt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AnkaraYBU-URO-SU-02
Record Dates: First submitted 2021-07-26; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Erectile Dysfunction Due to Diseases Classified Elsewhere; Covid19
Keywords: Erectile Dysfunction; COVID-19; Electromyography
MeSH Terms: conditions — COVID-19; Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: Corpus cavernosum electromyography, penile color Doppler ultrasonography and hormonal examinations were compared between the groups of patients with erectile dysfunction who did not have COVID-19, who were diagnosed with COVID-19 and were treated as outpatients or inpatients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients that had COVID-19 and were treated as outpatients (Active Comparator): Patients underwent diagnostic evaluation including IIEF-5 form, penile color Doppler ultrasonography, corpus cavernosum electromyography, and fasting serum levels of testosterone, luteinizing hormone, follicle stimulating hormone, and prolactin measured in the morning (07-11 am). The relaxation degrees of cavernosal smooth muscles were calculated from the corpus cavernosum electromyography results.
  Interventions: Diagnostic Test: corpus cavernosum electromyography
- Patients who were hospitalized due to COVID-19 (Active Comparator): Patients underwent diagnostic evaluation including IIEF-5 form, penile color Doppler ultrasonography, corpus cavernosum electromyography, and fasting serum levels of testosterone, luteinizing hormone, follicle stimulating hormone, and prolactin measured in the morning (07-11 am). The relaxation degrees of cavernosal smooth muscles were calculated from the corpus cavernosum electromyography results.
  Interventions: Diagnostic Test: corpus cavernosum electromyography
- Patients who did not have COVID-19 (Active Comparator): Patients underwent diagnostic evaluation including IIEF-5 form, penile color Doppler ultrasonography, corpus cavernosum electromyography, and fasting serum levels of testosterone, luteinizing hormone, follicle stimulating hormone, and prolactin measured in the morning (07-11 am). The relaxation degrees of cavernosal smooth muscles were calculated from the corpus cavernosum electromyography results.
  Interventions: Diagnostic Test: corpus cavernosum electromyography

INTERVENTIONS:
Diagnostic Test: corpus cavernosum electromyography — Cc-EMG was performed by using the cc-EMG module of Ellipse 4 device (Andromeda, Germany), which comprises of a 2-channel electromyography amplifier with a row sampling rate of 16 kHz, filtered sampling rate of 166.67 Hz and a band width of 0.5-30 Hz with the speed of the thermo-writer paper set at 5 mm/s. Measurements of the electrical activity of the corpus cavernosum (EACC) were done for 10 minutes using coaxial needle electrodes during the flaccid state and after intracavernous papaverine (60 mg) injection.

SUMMARY:
The aim of the study is to illuminate the role of COVID-19 in the pathophysiology of erectile dysfunction (ED). Nine patients that had COVID-19 and were treated as outpatients were classified as group 1, 10 patients who were hospitalized due to COVID-19 were classified as group 2, and 10 patients who did not have COVID-19 and applied to the urology outpatient clinic with ED complaints and had similar clinical characteristics were classified as the control group (group 3). Patients underwent diagnostic evaluation including International Index of Erectile Function-5 form, penile color Doppler ultrasonography, corpus cavernosum electromyography, and fasting serum levels of reproductive hormones (07-11 am). According to the results of our study, cavernous smooth muscle damage occurs in patients with COVID-19 and it has an important role in the pathophysiology of erectile dysfunction.

DETAILED DESCRIPTION:
COVID-19, which is caused by a novel coronavirus Sars-Cov-2, has been affecting people all over the world for more than a year and has resulted in many deaths. It can affect almost every part of the body and cause diseases including anosmia, hypogonadism, myopathy, neuropathy, and vasculitis. Studies have reported that it may cause erectile dysfunction (ED), however, its role in the pathophysiology of ED has not yet been fully elucidated.

Patients aged 20-50 years who applied to the urology outpatient clinic due to ED were included in the study. Nine patients that had COVID-19 and were treated as outpatients were classified as group 1, 10 patients who were hospitalized due to COVID-19 were classified as group 2, and 10 patients who did not have COVID-19 and applied to the urology outpatient clinic with ED complaints and had similar clinical characteristics were classified as the control group (group 3). Patients underwent diagnostic evaluation including International Index of Erectile Function (IIEF)-5 form, penile color Doppler ultrasonography (CDUS), corpus cavernosum electromyography (cc-EMG), and fasting serum levels of reproductive hormones (07-11 am).

According to penile CDUS results, distribution of vasculogenic pathologies in groups was as follows: 33% in group 1, 40% in group 2, and 40% in group 3. According to cc-EMG results, the pre-vasoactive drug (VAD) amplitudes of the patients in group 2 were significantly lower than those in group 3 (p: 0.005). Moreover, the pre-VAD amplitudes of the patients in group 1 were also significantly lower than those in group 3 (p: 0.042). In addition, while the RD values of the patients in group 2 were significantly lower than those in group 3, no significant difference was observed between other groups. There was no significant difference between the groups in terms of hormonal profile.

Cavernosal smooth muscle damage that occurs due to COVID-19-related endothelial dysfunction may disrupt the nutrition of cavernosal tissues. The deterioration of the nutrition of the cavernosal tissues may be one of the important reasons for the post-COVID-19 ED. The results of our study need to be confirmed with larger studies in which electromyographic as well as histopathological examinations are performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-50 years
* Applied to the urology outpatient clinic with the complaint of erectile dysfunction
* International Index of Erectile Function-5 score of <17

Exclusion Criteria:

* Patients with concomitant neurological disease
* Diabetes, coronary artery disease, kidney failure, hyperlipidemia, hypertension
* Smoking and alcohol addiction
* Hormonal drug use
* History of pelvic trauma and history of penile, testicular, pelvic or perineal surgery
* Diagnosis of malignancy
* Patients that used opioids within the last 3 months

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2021-02-20 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Corpus cavernosum electromyography amplitudes and frequency | 1 hour
  Measurements of the electrical activity of the corpus cavernosum were done for 10 minutes using coaxial needle electrodes during the flaccid state and after intracavernous papaverine (60 mg) injection
Corpus cavernosum electromyography relaxation degree | 1 hour
  Relaxation degree (RD) was defined as the percent decrease in the amplitudes of electrical activity of the corpus cavernosum(EACC). It can be formulated as RD = pre-injectional EACC (amp) - post-injectional EACC (amp) × 100/pre-injectional EACC (amp)

CONTACTS AND LOCATIONS:
Overall Officials: Onder Kayigil, Professor, Study Chair — Ankara Yildirim Beyazit University School of Medicine
Locations (1):
- Ankara Yildirim Beyazit University, Schhol of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Unal S, Uzundal H, Soydas T, Kutluhan MA, Ozayar A, Okulu E, Kayigil O. A possible mechanism of erectile dysfunction in coronavirus disease-19: Cavernosal smooth muscle damage: A pilot study. Rev Int Androl. 2023 Oct-Dec;21(4):100366. doi: 10.1016/j.androl.2023.100366. Epub 2023 Jun 13. PMID 37413939